CLINICAL TRIAL: NCT03642275
Title: iCardia4HF: A Patient-centered Mobile Health Intervention to Promote Self-care and Improve Patient Outcomes in Chronic Heart Failure
Brief Title: Patient-centered Mobile Health Intervention to Improve Self-care in Patients With Chronic Heart Failure
Acronym: iCardia4HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Spyros Kitsiou, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-0307
Record Dates: First submitted 2018-06-15; First posted 2018-08-22 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure
Keywords: heart failure; mHealth; smartphone; wearable electronic devices; text messaging; self-management; self-care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to patients' randomization assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iCardia4HF (Experimental): Participants will be using a heart failure mobile app, wearable activity tracking device, Bluetooth-enabled blood pressure monitor and weight scale for self-monitoring, and receive tailored text-messages about self-care.
  Interventions: Behavioral: iCardia4HF
- Control Group (No Intervention): Participants assigned to the usual care group will receive standard medical care, which includes nurse-led patient education about HF self-care before discharge, and follow-up visits at the UI Health, outpatient Heart Failure program.

INTERVENTIONS:
Behavioral: iCardia4HF — Participants in the intervention group will receive the Heart Failure Health Storylines mobile app, three connected health devices that interface with the app (Fitbit Charge 2 activity tracker, and FDA-approved Nokia BP monitor and Cardio Body weight scale), and a program of tailored self-care text-messages, in addition to usual care. Participants will be asked to use the app and devices to record and self-monitor their daily symptoms, blood pressure, weight, and physical activity.
  Arms: iCardia4HF

SUMMARY:
Approximately 6.5 million people have heart failure (HF) in the United States, and 960,000 new cases are reported each year. HF is one of the most common hospital diagnosis among older adults. About 40% of patients are readmitted within 1-year following their first admission for HF and hospitalization accounts for approximately 80% of the costs of HF management. This pilot study aims to assess the feasibility, acceptability, and preliminary efficacy of a patient-centered mobile health (mHealth) technology intervention in older adults with chronic heart failure.

DETAILED DESCRIPTION:
This is a single site, two-arm, pilot randomized controlled trial that aims to examine the feasibility, acceptability and preliminary efficacy of a mobile phone-based intervention compared to usual care in older adult patients with HF (≥50 years). Forty (n=40) patients from the University of Illinois Hospital & Health Sciences system will be enrolled in the study, randomly assigned to the intervention or usual care group, and followed for 60 days. Patients in the intervention group will receive the Heart Failure Health Storylines mobile app developed by Self Care Catalysts in collaboration with the Heart Failure Society of America, three connected health devices from Fitbit and Nokia that interface with the mobile app, and tailored text-messages targeting health beliefs, self-care efficacy, and knowledge about HF. The control group will receive standard care which involves patient education and outpatient follow up with physical and laboratory examinations as needed. The primary study outcome is change in self-care and quality of life. Secondary outcomes include hospital re-admissions and emergency room visits.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients or outpatients with a diagnosis of HF as defined by the International Classification of Diseases (ICD-10) codes
* Stage C, NYHA I, II or III
* ≥ 40 years of age
* Own a smartphone with text-messaging and internet plan
* Ability to speak and read English
* Live within 30 miles from UI Health

Exclusion Criteria:

* On an active waiting list for implanted ventricular assist device or heart transplant
* Advanced renal disease (dialysis or creatinine >4.0mg/dL)
* End-stage HF (hospice candidate)
* Active cancer
* Individuals who are not their own primary caregiver
* Discharge to a setting other than home
* Patients with baseline Montreal Cognitive Assessment (MoCA) score of < 22

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Self-care at 30 and 60 days | Baseline, 30 and 60 days
  Self-care will be measured with the Self-Care Heart Failure Index (SCHFI) v.6.2,87 which includes 3 subscales: self-care maintenance (10-items), self-care confidence (6-items), and self-care management (6-items). Standardized scores in each scale range from 0 to 100. A total score of ≥70 indicates adequate self-care.
Change from Baseline in Health-related Quality of Life (HRQoL) at 30 and 60 days | Baseline, 30 and 60 days
  HRQoL will be measured with the Kansas City Cardiomyopathy Questionnaire (23-items) that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Lower scores indicate worse HRQoL.

SECONDARY OUTCOMES:
Hospitalizations | 60 days
  The number of hospitalizations during the study will be measured with both self-report and the electronic medical record.
ER visits | 60 days
  The number of emergency room visits will be collected based on both self-reports and the electronic medical record

CONTACTS AND LOCATIONS:
Overall Officials: Spyros Kitsiou, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Hospital & Health Sciences System, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kitsiou S, Gerber BS, Buchholz SW, Kansal MM, Sun J, Pressler SJ. Patient-Centered mHealth Intervention to Improve Self-Care in Patients With Chronic Heart Failure: Phase 1 Randomized Controlled Trial. J Med Internet Res. 2025 Jan 15;27:e55586. doi: 10.2196/55586. PMID 39813671